CLINICAL TRIAL: NCT06130787
Title: Value of Biological Age, in Addition to Individual Frailty, for Personalising the Management of Cancer Treated with Targeted Therapy: the Model of Chronic Myeloid Leukemia Treated with Tyrosine Kinase Inhibitors.
Brief Title: Value of Biological Age, in Addition to Individual Frailty, for Personalising the Management of Cancer Treated with Targeted Therapy
Acronym: BIO-TIMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2023 BERGER; 2023-A00974-41 (Other: ANSM)
Record Dates: First submitted 2023-09-29; First posted 2023-11-14 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Leukemia,Myeloid, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental)
  Interventions: Biological: Blood and bone marrow sample

INTERVENTIONS:
Biological: Blood and bone marrow sample — Individual biological aging determined by DNA methylation analysis will be assessed at D0, M3 and M12.
  An optional bone marrow sample will be taken during the myelogram performed at diagnosis.
  Individual fragility and quality of life will be assessed using geriatric tools at D0, M6, M12, M24 and M36

SUMMARY:
French prospective multicenter, open-label study involving newly diagnosed CML patients. Two assessments will be performed during the follow-up of these patients: individual frailty using geriatric tools and individual biological aging determined by DNA methylation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* CML in chronic phase at time of diagnosis. Diagnosis must be made no more than 3 months (90 days) prior to inclusion. Diagnosis of chronic-phase CML (European Leukemia Network [ELN] 2020 criteria; Baccarani et al 2013) with confirmation of a Philadelphia chromosome (Ph1). A cryptic Ph1 chromosome must be confirmed by FISH.Criteria must meet the definition of chronic phase CML
* BCR ::ABL1 transcript quantifiable by quantitative PCR
* 1st-line treatment with tyrosine kinase inhibitor
* No tyrosine kinase inhibitor or hydroxyurea treatment received prior to first blood sampling (at diagnosis)
* Signature of informed consent for CML Observatory and signature of informed consent for BIO-TIMER protocol
* Read and understand French
* Enrolled in a social security plan or beneficiary of such a plan

Exclusion Criteria:

* CML in accelerated or blast phase
* Refusal to participate in the study
* Treatment started prior to inclusion
* Patients under guardianship, curatorship, deprivation of liberty or safeguard of justice
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2028-11-17 (Estimated)

PRIMARY OUTCOMES:
Biological age determination | Day 0;Month 3;Month 12
  The difference between biological age and chronological age (of the clone and the patient) expressed as a difference and as a percentage.
Individual fragility assessment | Day 0;Month 6;Month 12;Month 24;Month 36
  Individual fragility assessed by Geriatric Core Data set assessing social status, independence at home, mobility, nutrition, cognitive status, mood and comorbidities.
Individual fragility assessment | Day 0;Month 6;Month 12;Month 24;Month 36
  Individual fragility assessed by Rockwood clinical frailty score ranging from 1 (very fit) to 9 (at the end of life)
Tolerance of tyrosine kinase inhibitors | Day 0;Month 3;Month 6;Month 12;Month 24;Month 36
  Tolerance assessed by actual dose received
Tolerance of tyrosine kinase inhibitors | Day 0;Month 3;Month 6;Month 12;Month 24;Month 36
  Tolerance assessed by the number of tyrosine kinase inhibitor discontinuation due to intolerance
Tolerance of tyrosine kinase inhibitors | Day 0;Month 3;Month 6;Month 12;Month 24;Month 36
  Tolerance assessed by a description of adverse events as assessed by CTCAE v5.0
Tolerance of tyrosine kinase inhibitors | Day 0;Month 3;Month 6;Month 12;Month 24;Month 36
  Tolerance assessed by changes and number of tyrosine kinase inhibitor lines
Tolerance of tyrosine kinase inhibitors | Day 0;Month 3;Month 6;Month 12;Month 24;Month 36
  Tolerance assessed by a description of treatment sequences

SECONDARY OUTCOMES:
Distribution of individual clinical fragility levels assessed by Geriatric Core Data set at the time of diagnosis. | Day 0
  Individual fragility assessed by Geriatric Core Data set assessing social status, independence at home, mobility, nutrition, cognitive status, mood and comorbidities at the time of diagnosis.
Distribution of individual clinical fragility levels assessed by Rockwood clinical frailty score at the time of diagnosis. | Day 0
  Individual fragility assessed by Rockwood clinical frailty score ranging from 1 (very fit) to 9 (at the end of life) at the time of diagnosis.
Evaluation of therapeutic response through quantification of the BCR::ABL transcript | Month 3;Month 6;Month 12;Month 15;Month 18;Month 21;Month 24;Month 27;Month 30;Month 33;Month 36
  Quantification of BCR::ABL transcript expressed as copy number relative to 100 copies of control gene transcripts
Assessment of therapeutic response by quantification of residual disease | Month 3;Month 6;Month 12;Month 15;Month 18;Month 21;Month 24;Month 27;Month 30;Month 33;Month 36
  Decrease in residual disease and achievement of MMR (≤0.1%), MR4 (≤0.01%), MR4.5 (≤0.032%), MR5 (≤0.001%) thresholds)
Assessment of patients' quality of life | Day 0;Month 6;Month 12;Month 24;Month 36
  Quality of life assessed using the European Organisation for Research and Treatment of Cancer LG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients, with a higher score indicating a better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marc BERGER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (17):
- France (17):
  - CHU Annecy-Genevois, Annecy
  - Institut Bergonié, Bordeaux
  - CHU Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Créteil, Créteil
  - CHU Grenoble Alpes, Grenoble
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU Nancy, Nancy
  - Groupe Hospitalier Paris Saclay - Site de Bicêtre, Paris
  - CHU Rennes, Rennes
  - CHU Saint-Etienne, Saint-Etienne
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - CHU Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casile M, Albrand G, Lahaye C, Lebecque B, Besombes J, Bourgne C, Pereira B, Saugues S, Jamot C, Hermet E, Berger MG. Value of combining biological age with assessment of individual frailty to optimize management of cancer treated with targeted therapies: model of chronic myeloid leukemia treated with tyrosine kinase inhibitors (BIO-TIMER trial). BMC Cancer. 2024 May 30;24(1):661. doi: 10.1186/s12885-024-12415-2. PMID 38816821